CLINICAL TRIAL: NCT02547454
Title: Investigating the Effectiveness of Renal Anaemia Treatment in Pre-Dialysis Patients With Mircera in Daily Clinical Practice - MIRVITA
Brief Title: An Observational Study to Evaluate the Effectiveness of Mircera Treatment for Renal Anemia in Pre-dialysis Participants With Chronic Kideny Disease (CKD)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22069
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CKD participants treated with Mircera: Participants with CKD received Mircera, as per routine clinical practice and was followed for approximately 36 months.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta
  Other Names: Mircera

SUMMARY:
This observational trial will examine the efficacy and safety of Mircera for renal anemia in participants with stage III-IV CKD in daily clinical practice. Mircera will be prescribed by treating physician and followed for approximately 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged > 18 years with CKD
* Participants who are eligible for Mircera treatment according to current guidelines and summary of product characteristics (SmPC)

Exclusion Criteria:

* Non-renal anemia
* Pregnancy and breast-feeding
* Uncontrolled hypertension
* Known hypersensitivity to methoxy polyethylene glycol-epoetin beta
* Administration of any other study drug within 30 days prior to study enrollment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CKD who do not require dialysis and are appropriate for treatment with Mircera according to European Best Practice Guidelines (EBPG) and Kidney Disease Outcomes Quality Initiative (K/DOQI) guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2008-12-31 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Slovenia (12):
  - Hospital Celje; Dept For Kidney Disease & Dialysis, Celje
  - Splosna Bolnisnica Izola; Oddelek Za Nefrologijo, Izola
  - Clinical Centre Ljubljana; Clinical Dep. For Nephrology, Ljubljana
  - Nefroloska Ambulanta, Ljubljana
  - Hospital Maribor; Clinical Dept For Internal Medicine, Maribor
  - Splosna Bolnisnica Murska Sobota; Oddelek Za Nefrologijo, Murska Sobota
  - Zdravstveni Zavod Medicinski Center Šinigoj Nova Gorica, Nova Gorica
  - Hospital Novo Mesto; Dialysis Dept, Novo Mesto
  - Hospital Dr.Joze Potre; Dialysis Dept, Ptuj
  - Splosna Bolnisnica Franc Derganc; Oddelek Za Nefrologijo, Sempeter Pri Novi Gorici
  - Hospital Slovenj Gradec; Hemodialysis Dept, Slovenj Gradec
  - Splosna Bolnisnica Trbovlje; Oddelek Za Nefrologijo, Trbovlje

RESULTS

PARTICIPANT FLOW:
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants with chronic kidney disease (CKD), who did not require dialysis, received methoxy polyethylene glycol-epoetin beta (Mircera) either intravenously (IV) or subcutaneously (SC), as per routine clinical practice, and were followed for approximately 36 months.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Started | 393
Completed | 221
Not Completed | 172
Not completed — Due to hemodialysis | 53
Not completed — Due to transplantation | 1
Not completed — Due to no further need to treat | 4
Not completed — Death | 38
Not completed — Lost to Follow-up | 26
Not completed — Other | 39
Not completed — No data | 11

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants.
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants with CKD, who did not require dialysis, received methoxy polyethylene glycol-epoetin beta either IV or SC, as per routine clinical practice, and were followed for approximately 36 months.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216
  Male | 177

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hemoglobin (Hb) Value Within the Target Range (110 to 120 Grams Per Liter [g/L]) at Baseline
Description: If a participant had more than 1 assessment during the specified time frame, the last observed Hb value was considered for calculation.
Time Frame: Baseline
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 390
Percentage of participants | 22.8

2. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (110 to 120 g/L) at Months 1-3
Description: as for outcome 1
Time Frame: At Months 1-3
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 259
Percentage of participants | 34

3. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (110 to 120 g/L) at Months 4-6
Description: as for outcome 1
Time Frame: At Months 4-6
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 296
Percentage of participants | 35.1

4. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (110 to 120 g/L) at Months 7-9
Description: as for outcome 1
Time Frame: At Months 7-9
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 232
Percentage of participants | 32.3

5. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (110 to 120 g/L) at Months 10-12
Description: as for outcome 1
Time Frame: At Months 10-12
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 199
Percentage of participants | 35.2

6. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (110 to 120 g/L) at Months 13-15
Description: as for outcome 1
Time Frame: At Months 13-15
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 170
Percentage of participants | 33.5

7. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (110 to 120 g/L) at Months 16-18
Description: as for outcome 1
Time Frame: At Months 16-18
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 172
Percentage of participants | 31.4

8. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (110 to 120 g/L) at Months 19-21
Description: as for outcome 1
Time Frame: At Months 19-21
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 96
Percentage of participants | 26

9. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (110 to 120 g/L) After 21 Months up to 36 Months
Description: as for outcome 1
Time Frame: After 21 Months up to 36 Months
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 35
Percentage of participants | 31.4

10. Primary Outcome: Percentage of Participants With Hemoglobin (Hb) Value Within the Target Range (100 to 130 g/L) at Baseline
Description: as for outcome 1
Time Frame: At Baseline
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 390
Percentage of participants | 71.3

11. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (100 to 130 g/L) at Months 1-3
Description: as for outcome 1
Time Frame: At Months 1-3
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 259
Percentage of participants | 77.2

12. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (100 to 130 g/L) at Months 4-6
Description: as for outcome 1
Time Frame: At Months 4-6
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 296
Percentage of participants | 73.6

13. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (100 to 130 g/L) at Months 7-9
Description: as for outcome 1
Time Frame: At Months 7-9
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 232
Percentage of participants | 74.1

14. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (100 to 130 g/L) at Months 10-12
Description: as for outcome 1
Time Frame: At Months 10-12
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 199
Percentage of participants | 75.9

15. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (100 to 130 g/L) at Months 13-15
Description: as for outcome 1
Time Frame: At Months 13-15
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 170
Percentage of participants | 78.2

16. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (100 to 130 g/L) at Months 16-18
Description: as for outcome 1
Time Frame: At Months 16-18
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 172
Percentage of participants | 79.7

17. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (100 to 130 g/L) at Months 19-21
Description: as for outcome 1
Time Frame: At Months 19-21
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 96
Percentage of participants | 75

18. Primary Outcome: Percentage of Participants With Hb Value Within the Target Range (100 to 130 g/L) After 21 Months up to 36 Months
Description: as for outcome 1
Time Frame: After 21 Months up to 36 Months
Population: Analysis population included all enrolled participants who had at least one Hb assessment at the specified time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 35
Percentage of participants | 68.6

19. Secondary Outcome: Median Time in Which Hb Value Was Maintained Within Target Range of 110-120 g/L
Time Frame: Up to 36 Months
Population: Analysis population included all enrolled participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 390
Months | NA [NA to NA] — Median time (full range) to obtain Hb value within the target range was not possible to analyze due to fluctuation within and outside of range.

20. Secondary Outcome: Median Time in Which Hb Value Was Maintained Within Target Range of 100-130 g/L
Time Frame: Up to 36 Months
Population: Analysis population included all enrolled participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 393
Months | NA [NA to NA] — Median time (full range) to obtain Hb value within the target range was not analyzed due to fluctuation within and outside of range.

21. Secondary Outcome: Average Dose of Methoxy Polyethylene Glycol-Epoetin Beta
Description: Average dose of methoxy polyethylene glycol-epoetin beta administered at Baseline
Time Frame: Baseline
Population: Analysis population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: microgram
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 393
microgram | 88 (46)

22. Secondary Outcome: Median Dose of Methoxy Polyethylene Glycol-Epoetin Beta
Description: Median monthly dose of methoxy polyethylene glycol-epoetin beta administered in the study up to 36 months.
Time Frame: Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21 and After 21 Months up to 36 Months
Population: Analysis population included all enrolled participants. Here, n signifies participants with available data at specified time-point.
Measure: Median (Full Range); unit: microgram
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 393
microgram
  Month 1 (n=393) | 100 [50 to 400]
  Month 3 (n=263) | 75 [50 to 480]
  Month 6 (n=300) | 75 [30 to 300]
  Month 9 (n=239) | 67 [30 to 400]
  Month 12 (n=206) | 50 [25 to 360]
  Month 15 (n=175) | 50 [30 to 360]
  Month 18 (n=177) | 50 [30 to 250]
  Month 21 (n=93) | 50 [0 to 300]
  After 21 Months up to 36 Months (n=30) | 50 [30 to 250]

23. Secondary Outcome: Number of Dose Adaptations
Description: Total number of changes (increase or decrease) in daily methoxy polyethylene glycol-epoetin beta doses. The reasons for dose-adaptations included: inflammation or infection; kidney function decline; over-response; iron deficiency; insufficient response; adverse effect; start of maintenance dose; kidney function improvement; re-introduction of treatment; and others (other reasons than specified).
Time Frame: Up to 36 Months
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Events
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 393
Events
  Total dose adaptations | 729
  Inflammation or infection | 11
  Kidney function decline | 32
  Over response | 314
  Iron deficiency | 14
  Insufficient response | 213
  Adverse effect | 2
  Start of maintenance phase | 71
  Kidney function improvement | 4
  Re-introduction of treatment | 41
  Other | 27

24. Secondary Outcome: Percentage of Participants With Dose 0
Description: Percentage of participants who did not use methoxy polyethylene glycol-epoetin beta (Dose 0) at atleast one visit during study period.
Time Frame: Up to 36 Months
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 393
Percentage of participants | 32.6

25. Secondary Outcome: Percentage of Participants With Iron Replacement
Description: Iron replacement was given to the participants either in oral iron replacement or intravenous replacement or both.
Time Frame: Up to 36 Months
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 393
Percentage of participants
  Oral Iron Replacement | 37.7
  Intravenous Iron Replacment | 31.6
  Oral and Intravenous Iron Replacment | 10.9
  No Iron Replacment | 19.8

ADVERSE EVENTS:
Time Frame: Up to 36 Months
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Serious Adverse Events (participants affected / at risk) | 3/393
Other Adverse Events (participants affected / at risk) | 2/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=393)
Cerebrovascular accident (Nervous system disorders) | 1
Epileptic seizure (Nervous system disorders) | 1
Orthostatic collapse (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=393)
Rash (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.